CLINICAL TRIAL: NCT07155772
Title: Feasibility Study on a Prehospital Extracorporeal CardioPulmonary Resuscitation in the Pavia's Province. An Interventional Study on Complex Treatment Strategy
Brief Title: Feasibility Study on a Prehospital Extracorporeal CardioPulmonary Resuscitation in the Pavia's Province.
Acronym: eCPR on Site
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Alessandra Palo, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: eCPR on Site
Record Dates: First submitted 2025-08-07; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-02

CONDITIONS: Refractory Cardiac Arrest
Keywords: cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory cardiac arrest who receive extracorporeal cardiopulmonary resuscitation (Experimental)
  Interventions: Procedure: Extracorporeal CardioPulmonary Resuscitation (eCPR)

INTERVENTIONS:
Procedure: Extracorporeal CardioPulmonary Resuscitation (eCPR) — The intervention of this study consists of moving the current eCPR program out of the hospital to reduce the time from collapse to ECMO flow (low-flow time).

SUMMARY:
This is a single Center interventional study, assessing the feasibility of a complex treatment strategy where an in-hospital standard care process is applied in an out-of-hospital cardiac arrest.

The objective of this study is to investigate the feasibility of a prehospital eCPR program in the context of the Pavia province in order to reduce the time from cardiac arrest to organ reperfusion with thefarthest aim of improving survival and good neurologic outcomes of patient victims of refractory cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest occurred in Pavia province
* the age of the patient is between 18 and 70
* witnessed cardiac arrest
* CPR started within 5 minutes of the patient's collapse or presence of gasping at the arrival of the ACLS team
* eCPR team arrived within 60 minutes of the patient's collapse
* etCO2 ≥ 10 mmHg
* mechanical chest compression is ongoing
* refractory cardiac arrest after at least 15 minutes of ACLS

Exclusion Criteria:

* Modified Rankin Scale (mRS) ≥ 3
* Advanced COPD or other advanced pulmonary illness
* End-stage or metastatic neoplasm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
number of successful eCPR placed in prehospital settings over patients that meet inclusion criteria | up to 12 months
  Successful cannulation is described as maintaining an ECMO circulatory flow of 40 ml/kg/min or more for at least 5 minutes.

SECONDARY OUTCOMES:
Cause of cannulation failure | up to 12 months
Proportion of cannulation feasibility according to the implant site | up to 12 months
Evaluation of eCPR Team Performance | up to 12 months
  Evaluation of eCPR Team Performance to better design a definitive institutional eCPR program

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy